CLINICAL TRIAL: NCT06654011
Title: IN10018 Plus Nab-Paclitaxel and Cadonilimab for Metastatic, Recurrent, or Persistent Gastric-Type Adenocarcinoma of the Cervix: A Multicenter, Single-Arm, Phase II Trial
Brief Title: IN10018 With Nab-Paclitaxel and Cadonilimab for Metastatic or Recurrent Gastric-Type Cervical Adenocarcinoma: Phase 2 Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT240895
Record Dates: First submitted 2024-10-20; First posted 2024-10-23 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cervical Adenocarcinoma; Gastric-type Endocervical Adenocarcinoma
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): IN10018 is administered orally at a dose of 100 mg once daily; cadonilimab is given at a dose of 10 mg/kg via intravenous infusion on Day 1 of each cycle, every 3 weeks; and nab-paclitaxel is administered at a dose of 260 mg/m² via intravenous infusion on Day 1 of each cycle, also every 3 weeks. Patients will undergo a maximum of 6 cycles of this combination chemotherapy. Following this regimen, maintenance therapy will consist of a combination of cadonilimab and IN10018.
  Interventions: Drug: IN10018; Drug: Nab-paclitaxel; Drug: Cadonilimab

INTERVENTIONS:
Drug: IN10018 — 100 mg, orally, once daily
  Other Names: BI 853520
Drug: Nab-paclitaxel — 260 mg/m², IV infusion, Q3W
  Other Names: Albumin-bound paclitaxel
Drug: Cadonilimab — 10 mg/kg, IV infusion, Q3W
  Other Names: AK104

SUMMARY:
Gastric-type adenocarcinoma of the cervix is the most commonly diagnosed HPV-independent subtype of cervical cancer, characterized by a poor prognosis and limited responsiveness to existing therapies. Therefore, the exploration of new treatment modalities is critically important. This is an open-label, single-arm, multi-center clinical trial to evaluate the efficacy and safety of IN10018 plus nab-paclitaxel and cadonilimab in the treatment of adult women with metastatic, recurrent, or persistent gastric-type adenocarcinoma of the cervix.

DETAILED DESCRIPTION:
Subjects will receive IN10018 at a dose of 100 mg orally once daily, in combination with nab-paclitaxel at 260 mg/m² and cadonilimab at 10 mg/kg, both administered via intravenous infusion on Day 1 of each 3-week cycle. Tumor assessments will be conducted every 2 cycles throughout the treatment period. If the therapy proves effective, chemotherapy will continue for up to 6 cycles. Upon completion of chemotherapy, maintenance therapy with cadonilimab and IN10018 will begin and continue until either disease progression or the emergence of intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Females 18-75 years of age.
2. Patients must have metastatic, recurrent or persistent gastric-type adenocarcinoma of the cervix which is not amenable to curative treatment with surgery and/or radiation therapy.
3. Patients must have had at least one prior systemic chemotherapeutic regimen for metastatic, recurrent or persistent carcinoma of the cervix. (Note: Prior adjuvant therapy is NOT counted as a systemic chemotherapeutic regimen for management of metastatic, recurrent or persistent carcinoma of the cervix, adjuvant therapy includes cisplatin given concurrent with primary radiation therapy (CCRT).
4. Patients must have measurable disease per REClST 1.1; measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded as ≥ 10 mm with computed tomography (CT) scan, magnetic resonance imaging (MRI); a lymph node must be ≥ 15 mm in short axis.
5. Eastern Cooperative Oncology Group score 0-1.
6. Life expectancy exceeds 3 months.
7. AEs due to previous treatments should be resolved to ≤ Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy are eligible.
8. NEU ≥ 1.5*10^9 /L, Platelet ≥ 75×10^9 /L, Hemoglobin ≥ 90 g/L; Serum creatinine ≤ 1.5 times the upper limit of normal (ULN).; Urinary protein < 2+ or 24h urinary protein quantity < 1.0 g; AST and ALT ≤ 2.5 times ULN; Total bilirubin ≤ 1.5 times ULN; Albumin levels ≥ 28 g/L; Coagulation function: Prothrombin time (PT) and international normalized ratio (INR) ≤ 1.5 times the ULN.
9. Female participants must test negative for HCG in urine or blood, except in cases of menopause or prior hysterectomy. Female patients of childbearing potential and their partners must use effective contraception during the study and for 6 months after the final dose of the study drug.
10. Willing to participate in this study, and sign the informed consent.

Exclusion Criteria:

1. Patients with cervical cancer histologically diagnosed as squamous cell carcinoma, usual-type adenocarcinoma, clear cell carcinoma, adenosquamous carcinoma, small cell carcinoma, or any non-gastric-type adenocarcinoma.
2. Participate in other drug clinical trials at the same time.
3. Known hypersensitivity to any component of the IN10018 formulation or to cadonilimab.
4. Patients with active autoimmune disease or a history of autoimmune disorders.
5. Patients with concomitant conditions requiring immunosuppressive medications or systemic or absorbable local corticosteroids at immunosuppressive doses. The use of prednisone >10 mg/day or an equivalent dose is prohibited within 2 weeks prior to the first administration of the investigational drug.
6. HIV infection or a positive test for acquired immunodeficiency syndrome (AIDS).
7. Patients with a history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
8. Necrotic lesions identified within 4 weeks prior to enrollment, where there is a high risk of major bleeding as determined by the investigator.
9. Severe infections occurring within 4 weeks prior to the first dose of study treatment.
10. Known active tuberculosis (TB) or suspicion of active TB.
11. Untreated chronic hepatitis B infection or hepatitis B virus (HBV) carriers with HBV DNA levels exceeding 1000 IU/mL, or patients with active hepatitis C infection.
12. Patients with known leptomeningeal disease, spinal cord compression, or active brain metastases.
13. Uncontrolled severe medical conditions that, in the investigator's judgment, would interfere with the patient's ability to receive study treatment, including but not limited to severe cardiovascular disease, cerebrovascular disease, uncontrolled diabetes, or uncontrolled infections.
14. Receipt of a live vaccine within 4 weeks prior to the first dose of study treatment. Note: Inactivated seasonal influenza vaccines are permitted.
15. Pregnant or breastfeeding female patients, or female patients of childbearing potential who refuse to use effective contraception.
16. Patients with symptomatic or unstable third-space fluid accumulations (e.g., pleural effusion, ascites, pericardial effusion) requiring repeated drainage.
17. Patients with a prior genetic test report indicating mutations associated with hyperprogression under immunotherapy, such as MDM2/4 amplification or EGFR mutations.
18. Not eligible for the study judged by researchers.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Every 6 weeks from the time of the first dose of the study drug until the completion of treatment, lasting approximately 18 weeks.
  ORR is defined as the percentage of the participants in the ITT population who have a complete response (CR) or partial response (PR). The ORR will be assessed by a blind independent central reviewer per RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  PFS is defined as the time from the first dose of study treatment/randomization to the first documentation of disease progression or death due to any cause, whichever comes first
Disease Control Rate (DCR) | Every 6 weeks from the time of the first dose of the study drug until the completion of treatment, lasting approximately 18 weeks.
  DCR is defined as the proportion of patients who achieve complete response (CR), partial response (PR), or stable disease (SD) following treatment. The DCR will be assessed by a blind independent central reviewer per RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Peng Wu, Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China
Locations (2):
- China (2):
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei

IPD SHARING:
Plan to Share IPD: No
Ethical and legal considerations necessitate the protection of participants' privacy, particularly when dealing with sensitive data that may identify individuals. Additionally, if data analyses remain incomplete, disclosing individual participant data (IPD) could compromise the integrity of the results and lead to hasty conclusions.